CLINICAL TRIAL: NCT06898853
Title: The Effect of 0.1% Topical Ciclosporin A for 12-weeks on the Ocular Surface Innate and Adaptive Immune Response in Dry Eye Disease
Brief Title: The Effect of 0.1% Topical Ciclosporin A for 12-weeks on the Eye Surface Immune Cells in Dry Eyes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of New South Wales (Other)
Collaborators: University of Melbourne (Other)
Responsible Party: Principal Investigator, Soumen Sadhu, Coordinating Investigator, The University of New South Wales
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UNSW IIT Protocol 202412001
Record Dates: First submitted 2025-03-09; First posted 2025-03-27 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Dry Eye Disease (DED)
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: A single-center, examiner-blind, randomized, controlled clinical trial to evaluate and compare the effect of CsA 0.1% with its vehicle on the ocular surface EIC density, morphology, inflammatory markers and signs, symptoms in DED.
  Intervention: Subjects will be allocated randomly in a 1:1 ratio in one of the following groups.
  Group A - CsA 0.1% - Ikervis (CSL Seqirus, Parkville, Victoria) once daily at night-time + Cationorm (CSL Seqirus, Parkville, Victoria) four times daily in both eyes for 12-weeks.
  Group B - Cationorm (CSL Seqirus, Parkville, Victoria) four times daily in both eyes for 12-weeks.
  Follow-up period: 12-weeks
  Total study period: 14-weeks
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A - CsA 0.1% - Ikervis (CSL Seqirus, Parkville, Victoria) once daily at night-time + Cationorm (Experimental)
  Interventions: Drug: 0.1% Ciclosporin A eye drops; Drug: Mineral oils eye drops
- Group B - Cationorm (CSL Seqirus, Parkville, Victoria) four times daily in both eyes for 12-weeks. (Active Comparator)
  Interventions: Drug: Mineral oils eye drops

INTERVENTIONS:
Drug: 0.1% Ciclosporin A eye drops — The active intervention arm has CsA 0.1% - Ikervis (CSL Seqirus, Parkville, Victoria) and mineral oils lubricating eye drops - Cationorm (CSL Seqirus, Parkville, Victoria)
  Arms: Group A - CsA 0.1% - Ikervis (CSL Seqirus, Parkville, Victoria) once daily at night-time + Cationorm
Drug: Mineral oils eye drops — This arm is the comparator arm has mineral oils lubricating eye drops - Cationorm (CSL Seqirus, Parkville, Victoria)

SUMMARY:
Dry eye disease (DED) is a common, long-lasting condition that affects the surface of the eye. It happens when there's a problem with tear production or quality, which can lead to inflammation and discomfort. The immune system plays a big role in how DED develops and continues.

Researchers have found that in people with DED, there are more immune cells and inflammatory substances in the tears and on the eye's surface. This includes various types of immune cells, like T cells and dendritic cells, which are part of the body's defense system.

The first treatment for DED is usually artificial tears, but because the condition is chronic and can flare up, clinicians often use anti-inflammatory treatments too. One such treatment is cyclosporine A (CsA), which comes as eye drops. CsA works by reducing inflammation and affects how immune cells behave.

Researchers can study the immune cells on the eye's surface using a special microscopy technique called in vivo confocal microscopy (IVCM). A newer version of this method, called functional IVCM (Fun-IVCM), allows researchers to watch how these cells move and behave over time.

In the current study, researchers want to compare 0.1% CsA with a lubricating eye drop to see how they affect the immune cells on the eye's surface. The researchers will use Fun-IVCM to look at the number, shape, and movement of immune cells of the eye. The researchers will also collect samples from the eye's surface and tears to measure various markers of inflammation.

The goal is to better understand how CsA works in treating DED by directly observing its effects on the immune response in the eye, which is unexplored. This could help improve treatments for people suffering from this condition and expand the use of CsA in DED.

DETAILED DESCRIPTION:
The immune system plays a pivotal role in dry eye disease (DED) pathogenesis. An increased level of several tear cytokines, chemokines, expression of HLA-DR molecules and activation of antigen presenting cells - dendritic cells (DCs), and lymphocytes all plays a central role in DED pathogenesis . The increased expressions of CD4+ and CD8+ T cells in the ocular surface of DED patients suggest a potential role of adaptive immunity in DED chronicity. The presence of antigen-presenting cells in the ocular surface and the upregulation of MHC II, IL-2, IL-17, IL-6 and IFN- γ and other co-stimulatory molecules in the tears of DED patients indicates a possible activation of the local adaptive immune response.

The conjunctiva serves as a primary site for immunological and histochemical analysis in ocular surface diseases . Researchers have employed various techniques to study ocular surface immunology such as impression cytology, conjunctival biopsy and through real-time polymerase chain reaction, immunocytochemistry, and light microscopy. Flow cytometry is a powerful technique that allows for the phenotypic analysis of cells through immunolabeling of extracellular expressions of various immune cell markers. An increased expressions of activation markers like HLA-DR and various immune cell populations including T cells (CD3+, CD4+, and CD8+), B cells, natural killer cells, and monocytes (CD14+ cells) are observed in DED using flow cytometry on conjunctival impression cytology samples .

Historically, studying human ocular surface immune cells required invasive techniques. With the advent of in vivo confocal microscopy (IVCM), has enabled real-time, non-invasive visualization of ocular surface epithelial immune cells (EICs) and corneal nerves. Over the past 20 years, researchers have used IVCM to examine pathologic changes in various ocular surface disorders. It is evident from several IVCM studies that corneal EICs undergoes changes such as increase in density and changes in its morphology in all forms of DED. Conventional static IVCM captures section images at a single time point of the corneal EIC's, and their analysis is limited to its density and morphology. While the in vivo nature of IVCM prevents direct immune cell phenotyping, the observed cells are predominantly believed to be DCs based on their morphological characteristics. Therefore, the authors have used the term EICs to define immune cells density (EIC density) quantified using static-IVCM. Unlike this method, which limits identification of the immune cell type, a recently pioneered, novel technique called functional IVCM (Fun-IVCM) enables identification of the immune cell types in the cornea by observing their morphodynamics. This method involves capturing consecutive sequence and volume scan images over a 30-40-minute period, with intervals of 4-5 minutes. The images are then time-lapsed to identify dynamic behaviour of each immune cell. Based on their dynamic behaviour and morphology, cells can be differentiated into either epithelial T cells (highly motile, smaller body size) or dendritic cells (DC's, less motile, larger body size with dendrites). Anterior corneal stromal macrophages can also be identified. Time-lapsed images allow for the examination of additional cell motility parameters, such as instantaneous speed and displacement speed.

The first-line treatment for DED is artificial tears. But, due to the chronic nature of the disease and recurrent acute exacerbations anti-inflammatory therapies has been largely implemented. Consequently, many of the current therapeutic approaches target various inflammatory pathways, aiming to break the vicious cycle of DED. Both topical corticosteroids and immunosuppressants effectively reduce inflammation in DED. Topical corticosteroids are used in DED to control acute exacerbations of inflammation of the ocular surface, but their longer-term use is limited by their iatrogenic ocular side-effects. To contrast this, immunosuppressive agents such as ciclosporin A (CsA) have potential anti-inflammatory effect, with minimal local side-effects. The use of CsA in chronic DED can significantly reduce ocular surface staining, redness, inflammatory markers and improves dry eye symptoms. In brief, CsA dampens T cell proliferation by inhibiting the phosphatase calcineurin. CsA functions at different steps of the immune response, during antigen presentation and DC-T cell interaction. Innate immune cells are now seen as potentially important targets of CsA and may reflect simultaneous targeting of dendritic cells, macrophages, and neutrophils. In the ocular surface preliminary evidence suggest that CsA can significantly reduce activation markers such as HLA-DR, CD11c, certain apoptosis markers, and conjunctival T lymphocytes accompanied the clinical improvement in CsA-treated DED patients.

While a handful of clinical trials have evidenced the efficacy of CsA in reducing inflammation and improving symptoms of DED, the direct effect of CsA on ocular surface immune cells has not been studied in detail using static and using Fun-IVCM. Given the effect of CsA on both innate and adaptive immune cells, the authors hypothesise that the use of 0.1% CsA will have an inhibitory effect on the ocular surface immune response along with improvement of signs and symptoms of DED compared with its vehicle. This paper highlights the randomized clinical trial protocol to comprehensively study the effect of CsA on the ocular surface innate and adaptive immune system in DED. The study will investigate CsA's impact on DCs (CD11c+ DCs, HLA-DR), T helper cell populations (CD4+ T cells) through analysis of lymphocyte markers (CD45, CD3, CD4) and their associated cytokines (Th1 pathway cytokines), particularly IL-2, IFN- γ and IL-17 which is a primary target of CsA's immunomodulatory action.

1.2. Study aims and hypothesis Aim 1: To investigate and compare the effect of 12-weeks topical 0.1% CsA therapy on ocular surface innate and adaptive immune cells using imaging - Static-IVCM and Fun-IVCM (immune cell density, morphology and morphodynamic behaviours), immune cell phenotyping using conjunctival impression cytology and flow cytometry techniques and tear cytokine analysis (Multiplex bead assay assessing tear concentrations of IL-2, IL-4, IL-6, IL-12, IL-17, IL-23, IFN- γ) Hypothesis: CsA will have an inhibitory effect on the ocular surface innate and adaptive immune cell density, morphology and tear cytokines in DED.

Aim 2: To assess the association between DED signs, symptoms and immune cell characteristics and tear cytokines in DED Hypothesis: A direct relationship between immune cell characteristics, teat cytokines and DED signs, symptoms exist.

Aim 3: To investigate the temporal relationship between immune cell changes and clinical improvement Hypothesis: Changes in immune cell characteristics (density and dynamics) and inflammatory markers precede clinical improvement in signs and symptoms of DED following CsA treatment.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age and above
2. Participants should meet any two of the following DED diagnostic criteria: i) ocular surface disease index score of ≥23 and ii) Oxford staining score of ≥1 iii) Tear meniscus height < 0.2 mm.

Exclusion Criteria:

1. Participants currently using or with previous use of steroids, ciclosporin, lifitegrast or any anti-inflammatory eye drops in the last 6 months.
2. Participants with systemic CsA or tacrolimus
3. Known hypersensitivity or contraindication to the study medication or any of its ingredients.
4. Active intraocular inflammation.
5. Contact lens wear or the use of contact lenses in the last 4 weeks.
6. Active eye infections or history of critical illness.
7. DED secondary to Steven-Johnson syndrome and cicatricial conjunctival disease.
8. Participants with other ocular co-morbidities and medications for glaucoma.
9. Participants with previous history of ocular surgery in the past 6 months.
10. Any other active or inactive systemic condition, structural abnormality such as eyelid malposition's that in the judgment of the investigator could confound study assessments or limit compliance.
11. Pregnant/breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Corneal epithelial immune cell density | Baseline, 4-weeks, and 12-weeks
  Evaluation of change in corneal epithelial immune cell density using in vivo confocal microscopy. The outcome will be measured as the number of immune cells per square millimeter (cells/mm²) of corneal epithelium. Higher values indicate increased immune cell infiltration and greater corneal inflammation.
Conjunctival immune cell density | Baseline, 4-weeks and 12-weeks.
  Evaluation of change in conjunctival immune cell density using impression cytology and flow cytometry. The outcome will be measured as the percentage change in specific immune cell populations (including CD45, CD3, CD4, CD8, CD11c, and HLA-DR positive cells). Higher percentage indicates an increase in immune cell density.

SECONDARY OUTCOMES:
Tear cytokine concentrations | Baseline and 12-weeks.
  Evaluation of change in tear film inflammation through measurement of cytokine concentrations in tear fluid. The concentration of each inflammatory cytokine (IL-2, IL-4, IL-6, IL-12, IL-17, IL-23, IFN-γ) will be individually measured and reported in picograms per milliliter (pg/mL). Higher concentrations indicate more severe ocular surface inflammation.
Tear film break-up time | Baseline, 4-weeks, and 12-weeks.
  Evaluation of change in tear-film break-up time observed through slit-lamp biomicroscopy after fluorescein dye instillation in the eye. The measurement is recorded in seconds, with lower values indicating decreased tear film stability and more severe dry eye disease. A value of <10 seconds is considered abnormal
Ocular surface disease index score | Baseline, 4-weeks and 12-weeks.
  Evaluation of change in dry eye symptoms using the Ocular Surface Disease Index (OSDI) questionnaire. The OSDI is a validated 12-item questionnaire that assesses symptoms related to dry eye disease and their impact on vision-related functioning. The scale ranges from 0 to 100 points, with higher scores indicating more severe dry eye symptoms
Ocular surface staining score | Baseline, 4-weeks and 12-weeks.
  Evaluation of change in ocular surface staining score using the Oxford Staining grading. The Oxford Staining Score is a standardized grading system that quantifies corneal and conjunctival epithelial damage by assessing the degree of fluorescein and/or lissamine green staining. The scale ranges from 0 to 5 points (or grades), with higher scores indicating more severe ocular surface damage.

CONTACTS AND LOCATIONS:
Overall Officials: Fiona Stapleton Professor, PhD, Principal Investigator — The University of New South Wales
Locations (1):
- School of Optometry and Vision Science, Sudney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Undecided